CLINICAL TRIAL: NCT00060268
Title: A Phase I/II Trial for Treatment of Obstructive Esophageal Tumors by Photodynamic Therapy (PDT) Using 2-(1-Hydroxyethyl)-2-Devinylpyropheophorbide-a (HPPH)
Brief Title: Photodynamic Therapy Using HPPH in Treating Patients With Obstructive Esophageal Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Hector Nava, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000301589; RPCI-DS-9701
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Esophageal Cancer
Keywords: recurrent esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: HPPH — iv

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make tumor cells more sensitive to light to kill tumor cells. Photosensitizing drugs such as HPPH are absorbed by tumor cells and, when exposed to light, become active and kill the tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of photodynamic therapy with HPPH in treating patients who have obstructive esophageal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine, preliminarily, the safety of HPPH in patients with obstructive esophageal tumors undergoing photodynamic therapy.
* Determine, preliminarily, tumor response in patients treated with this drug.
* Determine the length of time for cutaneous photosensitivity at the various drug doses in these patients.
* Determine plasma clearance rates for this drug in these patients.

OUTLINE: This is a dose-escalation study.

* Phase I: Patients receive HPPH IV over 1 hour on day 1. Patients then undergo laser light therapy on day 2.

Cohorts of 3 patients receive escalating doses of HPPH and a single light dose until the optimal dose is determined. The optimal dose is defined as the minimum dose producing efficacy without unacceptable toxicity.

* Phase II: Patients receive treatment as in phase I at the optimal dose. Patients are followed monthly for 6-24 months.

PROJECTED ACCRUAL: A total of 9-14 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal cancer

  * Stages T1-T3, any N, any M
* Tumor partially or completely obstructing the esophagus
* Primary or recurrent tumor meeting 1 of the following criteria for treatment:

  * Patient is too debilitated for or refused conventional therapy
  * Recurred after or failed to respond to chemotherapy, radiotherapy, or surgery
  * Deemed most appropriately treated by photodynamic therapy (PDT) in the opinion of the physician
* Persistent symptomatic disease required in patients who received prior radiotherapy, chemotherapy, or PDT with photofrin or HPPH

  * Prior PDT with HPPH allowed only if tumor is evident outside of the original treatment site
* No tracheal or bronchial involvement by bronchoscopy
* No T4 lesions involving the aorta, lung, or pericardium by CT scan, MRI, or endoscopic ultrasonography

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic

* Bilirubin no greater than 3.0 mg/dL
* Alkaline phosphatase no greater than 3 times upper limit of normal (ULN)
* SGOT no greater than 3 times ULN
* PT no greater than 1.5 times ULN

Renal

* Creatinine no greater than 3.0 mg/dL

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No contraindications to endoscopy
* No porphyria
* No hypersensitivity to porphyrins

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No concurrent photosensitizing agents (e.g., tetracyclines, sulfonamides, phenothiazines, sulfonylureas, hypoglycemic agents, thiazide diuretics, and griseofulvin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1997-01; Primary Completion 2003-09 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector R. Nava, MD, FACS, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States